CLINICAL TRIAL: NCT02998060
Title: Clinical Evidence of Robot Guided vs. Navigated vs. Free Hand Lumbar Spinal Fusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design [Randomization not feasible]
Sponsor: Marc Schröder (Other)
Responsible Party: Sponsor-Investigator, Marc Schröder, MD, PhD, Bergman Clinics
Organization: Bergman Clinics (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABR-59636
Record Dates: First submitted 2016-12-11; First posted 2016-12-20 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Spondylolisthesis; Intervertebral Disc Degeneration
Keywords: Robot; Spinal Fusion; Spine; Navigation; Freehand
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Robot-guided (Active Comparator): Robotic guidance (SpineAssist®or Renaissance® (Mazor Robotics Ltd. Caesarea, Israel) will be used for navigation and insertion of pedicle screws.
  Interventions: Procedure: Pedicle Screw Placement; Device: SpineAssist®/Renaissance® (Mazor Robotics Ltd. Caesarea, Israel)
- Navigated (Active Comparator): A computer-assisted method of navigation (CT- or 3D-Fluoroscopy-based) will be used for navigation and insertion of pedicle screws.
  Interventions: Procedure: Pedicle Screw Placement; Device: 3D C-Arm (Ziehm Imaging, Nuremberg, Germany)
- Freehand (Active Comparator): Pedicle screws will be inserted using the freehand technique under fluoroscopic control.
  Interventions: Procedure: Pedicle Screw Placement

INTERVENTIONS:
Procedure: Pedicle Screw Placement — As a part of the lumbar spinal fusion procedure, posterior pedicle screws will be placed.
Device: SpineAssist®/Renaissance® (Mazor Robotics Ltd. Caesarea, Israel) — This robot will be used to guide pedicle screws into their trajectories.
  Arms: Robot-guided
Device: 3D C-Arm (Ziehm Imaging, Nuremberg, Germany) — This 3D Fluoroscope will be used to navigate pedicle screws into their trajectories.
  Arms: Navigated

SUMMARY:
Computer-based navigation systems were first introduced to spine surgery in 1995 and while they have been long established as standards in certain cranial procedures, they have not been similarly adopted in spine surgery. Designed to overcome some of the limitations of navigation-based technologies, robot-guided surgical systems have become commercially available to surgeons worldwide.These systems are rapidly challenging the gold standards.

The aim is to conduct a prospective randomized controlled trial. The randomized variable will be the screw placement technique used. One arm will be treated with lumbar fusion using robotic guidance (RG), one arm will receive the same procedure but with a free hand technique (FH) and the third arm will use navigation (NV) (CT or Fluoroscopy-assisted). Intraoperative screw revisions and revision surgery for screw malposition as well as clinical patient-reported outcomes to identify any such differences between these methods of screw insertion will be assessed.

DETAILED DESCRIPTION:
A decade ago, minimally invasive surgery (MIS) was considered a promising development in spine surgery, yet the value of the pioneering technologies was questionable. With the growing number of experienced MIS surgeons, the influx of evidence in favour of MIS is rapidly increasing. This makes a compelling argument towards MIS offering distinct clinical benefits over open approaches in terms of blood loss, length of stay, rehabilitation, cost-effectiveness and perioperative patient comfort. Due to the limited or inexistent line-of-sight in MIS procedures, surgeons need to rely on imaging, navigation, and guidance technologies to operate in a safe and efficient manner. Therefore, a plethora of new and ever improving navigational systems have been developed. These systems allow a consistent level of safety and accuracy, on par with results achieved by very experienced free hand surgeons, with a reasonably short learning curve.

Computer-based navigation systems were first introduced to spine surgery in 1995 and while they have been long established as standards in certain cranial procedures, they have not been similarly adopted in spine surgery. Designed to overcome some of the limitations of navigation-based technologies, robot-guided surgery has become commercially available to surgeons worldwide, like SpineAssist® (Mazor Robotics Ltd. Caesarea, Israel) and the recently launched ROSA™ Spine (Zimmer-Biomet, Warsaw, Indiana, USA). These systems are rapidly challenging the gold standards.

SpineAssist®, and its upgraded version, the Renaissance®, provides a stable drilling platform and restricts the surgeon's natural full range of motion to 2 degrees of freedom (up/down motion and yaw in the cannula). The system's guidance unit moves into the trajectory based on exact preoperative planning of pedicle screws, while accounting for changes in intervertebral relationships such as due to distraction, cage insertion or changes between the supine patient position in the preoperative CT and the prone patient on the operating table. Published evidence on robot-guided screw placement has demonstrated high levels of accuracy with most reports ranging around 98% of screws placed within the pedicle or with a cortical encroachment of less than 2 mm.

Although the reliability and accuracy of robot-guided spine surgery have been established, the actual benefits for the patient in terms of clinical outcomes and revision surgeries remain unknown.

The investigators recently conducted a cohort study that showed some evidence that robotic guidance lowers the rate of intraoperative screw revisions and implant related reoperations compared to free hand procedures, while achieving comparable clinical outcomes. Now, these factors, among others, have to be assessed on a higher level of evidence. This would be, to date, the first randomized controlled trial comparing clinical patient reported outcomes of robotic guided (RG) pedicle screw placement vs. navigated (NV) vs. free hand (FH) pedicle screw placement.

The investigator's aim is to conduct a prospective randomized controlled trial. The randomized variable will be the screw placement technique used. One arm will be treated with lumbar fusion using robotic guidance (RG), one arm will receive the same procedure but with a free hand technique (FH) and the third arm will use navigation (NV) (CT or Fluoroscopy-assisted).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Lumbar single level discopathy or Spondylolisthesis of Meyerding Grade 1 or 2
* Body Mass Index >19 and <33
* American Society of Anesthesiologists Scale 1 or 2

Exclusion Criteria:

* Severe Scoliosis (Coronal Cobb's >30 degrees / Schwab classification sagittal modifier + or ++)

Ages: 17 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Quality of Life after Spinal Fusion as assessed using the Euroqol EQ-5D questionnaire | 12 months after surgery
Back Pain after Spinal Fusion as assessed using the Oswestry Disability Index (ODI) | 12 months after surgery
Back and Leg pain after Spinal Fusion as assessed using a Virtual Analogue Scale (VAS) | 12 months after surgery

SECONDARY OUTCOMES:
Number of Pedicle Screws that needed intraoperative Revision | Intraoperatively (From induction until end of anesthesia)
  If a pedicle screw is malpositioned and this is noticed intraoperatively, the screw can be removed and revised.
Number of Revision Surgeries for malpositioned Screws | Through study completion, an average of 12 months
  If a screw malposition is not detected intraoperatively and neurological deficits or other complaints secondary to the malpositioned screw arise, the screw needs to be surgically revised.

CONTACTS AND LOCATIONS:
Overall Officials: Victor E Staartjes, Stud. Med., Principal Investigator — University of Zurich
Locations (2):
- Universitätsmedizin Göttingen Georg-August, Göttingen, Lower Saxony, Germany
- University Hospital Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No